CLINICAL TRIAL: NCT06210490
Title: A Clinical Study of the Efficacy and Safety of Disitamab Vedotin in Combination With Radiotherapy for the Adjuvant Treatment of HER2 Overexpressing UTUC Patients With High Risk Factors for Recurrence After Radical Surgery
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Peking University First Hospital (Other)
Collaborators: Peking University First Hospital Miyun Hospital (Unknown)
Responsible Party: Principal Investigator, Xuesong Li, Peking University First Hospital, Peking University First Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RCVDUCIIR013
Record Dates: First submitted 2024-01-03; First posted 2024-01-18 (Actual); Last update posted 2025-12-15 (Actual); Status verified 2025-12

CONDITIONS: Upper Urinary Tract Urothelial Carcinoma
MeSH Terms: interventions — disitamab vedotin; Radiotherapy; Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Adjuvant therapy group (Experimental)
  Interventions: Drug: Disitamab Vedotin; Radiation: Radiotherapy
- Non-adjuvant therapy group (Active Comparator)
  Interventions: Other: Standard of Care

INTERVENTIONS:
Drug: Disitamab Vedotin — Disitamab vedotin (RC48-ADC) is a novel humanized anti-human epidermal growth factor receptor 2 (HER2) antibody conjugated with monomethyl auristatin E via a cleavable linker. Two phase II studies, RC48-C005 (NCT03507166) and RC48-C009 (NCT03809013), have shown its significant antitumor potential in patients with la/mUC with HER2 overexpression (immunohistochemistry (IHC) 3+ or 2+). In 2022, RC48-ADC was approved for patients with HER2 overexpressing la/mUC who had received prior chemotherapy in China.
  Arms: Adjuvant therapy group
Radiation: Radiotherapy — Radiotherapy dose: 45-50 Gy/25f/5w to lymph node drainage area; 62.5 Gy/25f/5w to metastatic or suspected metastatic lymph nodes.
  Arms: Adjuvant therapy group
Other: Standard of Care — Standard of Care
  Arms: Non-adjuvant therapy group

SUMMARY:
In this study, 60 patients with HER2 overexpression UTUC with high-risk recurrence factors after radical surgery were proposed to be enrolled, and were assigned to Cohort I (receiving adjuvant therapy group) and Cohort II (refusing to receive adjuvant therapy group) according to the subjects' wishes. Cohort I subjects were treated with vedicloxacinumab in combination with radiotherapy, and vedicloxacinumab treatment lasted for 6 months. Cohort II subjects receive close observation and best supportive care. Safety evaluations and efficacy evaluations will be performed during the study period. Safety Evaluations: Safety evaluations will be conducted within 3 days prior to each dose and will continue until 30 days after the last study dose or initiation of new antitumor therapy for subjects who have received at least one dose of study drug. Evaluation of effectiveness: effectiveness evaluations will be conducted every 12 weeks (±3 days) until imaging-confirmed tumor recurrence, subject death, withdrawal of informed consent, loss to follow-up, or study termination, whichever occurs first. Tumor assessment was performed according to the Criteria for Evaluation of Efficacy in Solid Tumors (RECIST v1.1). For subjects with disease progression, postoperative tumor recurrence, or initiation of other antitumor therapy, survival follow-up was performed every 3 months (window period ± 14 days) from the date of notification to collect information on the subject's subsequent antitumor therapy and survival until the subject's death, withdrawal of informed consent, loss of visit, or study termination, whichever occurred first.

ELIGIBILITY:
Inclusion Criteria:

1. Voluntary enrollment and signing of written informed consent;
2. Age ≥ 18 years, male or female;
3. Pathologically confirmed UTUC with at least any one of the following conditions: ① pT2 (need to be combined with at least simultaneous G3/high-grade tumor multiple, multifocal positive margins and one of the high-risk recurrence factors); ② pT3 to pT4; ③ pN+;
4. Cisplatin intolerance or not receiving platinum-based drugs for adjuvant therapy;
5. No recurrent metastasis confirmed by imaging ≥4 weeks postoperatively;
6. HER2 immunohistochemistry (IHC) results of IHC 3+ or 2+, subject's previous test results (confirmed by the investigator), and study center results are acceptable;
7. Expected survival time ≥ 6 months;
8. Eastern Cooperative Oncology Group (ECOG) Physical Status (PS) score of 0 to 1;
9. Normal major organ function, i.e., fulfillment of the following criteria:

   * Routine blood tests (no blood transfusion and no G-CSF use within 14 days prior to screening): a) Hemoglobin ≥ 90 g/L; b) Absolute neutrophil count (ANC) ≥ 1.5 x 10^9/L; c) Leukocyte count ≥ 3.0 × 10^9 /L; d) Platelet count ≥ 80 × 10^9/L ②Blood biochemistry (no albumin use within 14 days prior to screening): a) Albumin ≥ 28 g/L; b) Total bilirubin ≤ 2 x upper limit of normal (ULN); c) Aspartate aminotransferase (AST), alanine aminotransferase (ALT), and alkaline phosphatase (ALP) ≤ 2.5 x ULN in the absence of liver metastases, and ALT, AST, and ALP ≤ 5 x ULN in the presence of liver metastases; d) Creatinine ≤ 1.5 x ULN or creatinine clearance (CrCl) ≥ 50 mL/min calculated by the Cockcroft-Gault formula ③Coagulation: a) International Normalized Ratio (INR) or Prothrombin Time (PT) ≤ 1.5 x ULN; b) Activated partial thromboplastin time (APTT) ≤ 1.5 × ULN.

Exclusion Criteria:

1. A history of malignancy other than uroepithelial carcinoma, except in the following two cases: a) The patient has received potentially curative therapy and has had no evidence of the disease for 5 years; b) Basal cell carcinoma of the skin, squamous cell carcinoma of the skin, superficial bladder cancer, carcinoma in situ of the uterine cervix, and other carcinomas in situ for which resection was successfully received;
2. Prior allogeneic stem cell or parenchymal organ transplantation;
3. Patients who have received other prior anti-tumor systemic therapy (including herbal medicine with anti-tumor indications) less than 4 weeks after completion of therapy and prior to dosing in this study, or who have not recovered from adverse events caused by prior therapy to ≤ CTCAE grade 1 (with the exception of alopecia and hyperpigmentation);
4. Prior or current congenital or acquired immunodeficiency disease;
5. Active or previously documented autoimmune or inflammatory diseases (including, but not limited to: autoimmune hepatitis, interstitial pneumonia, inflammatory bowel disease, systemic lupus erythematosus, vasculitis, uveitis, pituitary gland inflammation, hyper- or hypothyroidism, and asthma requiring bronchodilator therapy), with vitiligo, or asthma that has resolved completely in childhood and does not require any intervention in adulthood;
6. Treatment with systemic immunosuppressive medication within 2 weeks prior to enrollment or anticipated need for systemic immunosuppressive medication during the study period, with the exception of the following: a) Intranasal, inhaled, topical, or locally injected (e.g., intra-articular injection) corticosteroids; b) Systemic corticosteroids in doses not exceeding 10 mg/day of prednisone or other equivalent effect; c) Prophylactic corticosteroids for hypersensitivity reactions;
7. Patients with a known or suspected history of hypersensitivity to vedicilumab and similar drugs, or a history of hypersensitivity to chimeric or humanized antibodies or fusion proteins, or to excipients of the study drug;
8. Prior thrombosis or thromboembolic event within the previous 6 months, such as stroke and/or transient ischemic attack, deep vein thrombosis, pulmonary embolism, etc;
9. Patients assessed by a physician to be at risk for severe bleeding, including but not limited to severe bleeding (> 30 ml within 3 months), hemoptysis (> 5 ml within 4 weeks), with gastroscopy/assessment in the event of any of the above, whichever is based on the microscopic assessment or active bleeding or coagulation abnormality, with a propensity to hemorrhage or undergoing thrombolytic, anticoagulant, or antiplatelet therapy;
10. clinically significant cardiovascular disease including, but not limited to, acute myocardial infarction, severe/unstable angina or coronary artery bypass grafting within the previous 6 months, congestive heart failure (New York Heart Association NYHA classification > grade 2), arrhythmias that are poorly controlled or require pacemaker therapy, hypertension that is uncontrolled by medications (systolic blood pressure ≥ 140 mmHg and/or diastolic blood pressure ≥ 90 mmHg);
11. Other significant clinical and laboratory abnormalities that, in the opinion of the investigator, compromise the safety evaluation, e.g., uncontrolled diabetes mellitus, chronic kidney disease, grade II or greater peripheral neuropathy (CTCAE V5.0), abnormal thyroid function;
12. Serious infections that are active or poorly controlled clinically active infections, including: a) Positive for the AIDS virus (HIV) (HIV1/2 antibodies); b) Active Hepatitis B (HBsAg positive or HBV DNA > 2000 IU/ml and abnormal liver function); c) Active hepatitis C (HCV antibody positive or HCV RNA ≥103 copies/ml and abnormal liver function); d) Active tuberculosis; e) Other uncontrolled active infection (CTCAE V5.0 > grade 2);
13. Not yet recovered from surgery, e.g. presence of unhealed incisions or serious postoperative complications;
14. Women who are pregnant or breastfeeding, and female or male patients of childbearing potential who are unwilling or unable to use effective contraception;
15. other conditions that the investigator deems inappropriate for inclusion.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-02-20 (Actual); Primary Completion 2028-05-31 (Estimated); Study Completion 2028-05-31 (Estimated)

PRIMARY OUTCOMES:
Disease Free Survival (DFS) | Follow-up every 12 weeks ± 7 days, for approximately 2 years

SECONDARY OUTCOMES:
Overall Survival (OS) | Follow-up every 12 weeks ± 7 days, for approximately 2 years
Metastasis-Free Survival (MFS) | Follow-up every 12 weeks ± 7 days, for approximately 2 years
Local-Recurrence Free (LRF) | Follow-up every 12 weeks ± 7 days, for approximately 2 years
Over-time Changes in ECOG PS scores | Follow-up every 12 weeks ± 7 days, for approximately 2 years
  Ecog PS score
  Eastern Cooperative Oncology Group (ECOG) Performance Status: the minimum value is 0 and maximum value is 4. Higher scores mean a worse outcome.
Over-time Changes in tumor markers | Follow-up every 12 weeks ± 7 days, for approximately 2 years
Adverse events and serious adverse events | Follow-up every 12 weeks ± 7 days, for approximately 2 years

CONTACTS AND LOCATIONS:
Locations (1):
- Peking University First Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Sheng X, Yan X, Wang L, Shi Y, Yao X, Luo H, Shi B, Liu J, He Z, Yu G, Ying J, Han W, Hu C, Ling Y, Chi Z, Cui C, Si L, Fang J, Zhou A, Guo J. Open-label, Multicenter, Phase II Study of RC48-ADC, a HER2-Targeting Antibody-Drug Conjugate, in Patients with Locally Advanced or Metastatic Urothelial Carcinoma. Clin Cancer Res. 2021 Jan 1;27(1):43-51. doi: 10.1158/1078-0432.CCR-20-2488. Epub 2020 Oct 27. PMID 33109737
- [Background] Sheng X, Wang L, He Z, Shi Y, Luo H, Han W, Yao X, Shi B, Liu J, Hu C, Liu Z, Guo H, Yu G, Ji Z, Ying J, Ling Y, Yu S, Hu Y, Guo J, Fang J, Zhou A, Guo J. Efficacy and Safety of Disitamab Vedotin in Patients With Human Epidermal Growth Factor Receptor 2-Positive Locally Advanced or Metastatic Urothelial Carcinoma: A Combined Analysis of Two Phase II Clinical Trials. J Clin Oncol. 2024 Apr 20;42(12):1391-1402. doi: 10.1200/JCO.22.02912. Epub 2023 Nov 21. PMID 37988648